CLINICAL TRIAL: NCT03525665
Title: Study on the Role of FDG-PET in Patients With Follicular Lymphoma at Time of Relapse/Progression
Brief Title: Study on the Role of FDG-PET in Patients With FL at Time of Relapse/Progression
Status: Completed | Type: Observational
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Sponsor
Other Study IDs: FIL_PETRA
Record Dates: First submitted 2018-05-03; First posted 2018-05-16 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Follicular Lymphoma
Keywords: Follicular lymphoma; FDG-PET; Relapse/progression
MeSH Terms: conditions — Lymphoma, Follicular; Recurrence; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Metabolic activity measured by FDG-PET — To evaluate whether metabolic activity measured by FDG-PET (SUV max) at time of relapse is predictive of patient's outcome.

SUMMARY:
The study is designed as a retrospective analysis of patients with relapsed/refractory FL identified by the hematological centers of Italy.

DETAILED DESCRIPTION:
The study does not require any intervention on the patient, but it involves the simple collection of data that are already present in the medical record. Since this is a retrospective study, it will not require further analysis or diagnostic investigations than those already made.

ELIGIBILITY:
Inclusion Criteria:

* Patients with initial diagnosis of follicular lymphoma since 2001
* Histological confirmation of follicular lymphoma, grade I, II, III according to WHO 2008 classification, at the time of initial diagnosis
* Systemic first-line treatment with immuno-chemotherapy
* PET availability at the time of response after first-line treatment (optional)
* Clinical and radiological evidence of FL relapse or progression
* Histological confirmation of relapse (strongly recommended)
* PET availability of at the time of relapse/progression and images available for central assessment
* Availability of clinical, laboratory and therapeutic treatment data at the time of initial diagnosis and relapse/progression
* Follow up of at least 12 months after relapse/progression

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with relapsed/refractory FL identified by the hematological centers of Italy
Sampling Method: Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
PFS | 24 months
  Progression free survival from time of relapse/progression

SECONDARY OUTCOMES:
OS | 24 months
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Luminari, Principal Investigator — Ematologia - AO Arcispedale Santa Maria Nuova - IRCCS
Locations (27):
- Italy (27):
  - U.O.C. Ematologia Ospedale "San Nicola Pellegrino" ASL BAT, Trani, BT
  - Azienda Ospedaliera S. Gerardo Di Monza, Monza, Monza Brianza
  - CROB, Rionero in Vulture, Potenza
  - Università Cattolica del Sacro Cuore - Policlinico "A. Gemelli", Roma, RM
  - Emat Univ - Città della salute e della scienza di Torino, Torino, TO
  - SOS Ematologia Ospedale C. Massaia, Asti
  - A.O. Spedali Civili di Brescia - Ematologia, Brescia
  - Arnas Nuovo Ospedale Garibaldi Nesima - U.O.C. Ematologia, Catania
  - Az. Ospedaliero Universitaria Careggi, Florence
  - Divisione di Ematologia Ospedale Vito Fazzi, Lecce
  - AO Ospedale Civile di Legnano, Legnano
  - Ematologia Ospedale Madonna delle Grazie, Matera
  - Ospedale Ca' Granda-Niguarda, Milan
  - Policlinico di Modena - Università degli studi, Modena
  - AOU Maggiore della Carità di Novara - SCDU Ematologia, Novara
  - AOU Padova, Padua
  - Azienda Ospedaliera V.Cervello, Palermo
  - U.O. Ematologia e Centro Trapianto Midollo Osseo - Ospedale G. da Saliceto, Piacenza
  - A.O.R. "San Carlo" - U.O. Ematologia, Potenza
  - AO Bianchi Melacrino Morelli UO Ematologia, Reggio Calabria
  - AO Arcispedale S.Maria Nuova Ematologia, Reggio Emilia
  - Policlinico Universitario Campus Bio-Medico - "Area Ematologia Trapianto Cellule Staminali Medicina Trasfusionale e Terapia cellulare", Roma
  - Asl Ta Di Taranto, Taranto
  - Azienda Ospedaliera "S. Maria", Terni
  - A.O. C. Panico, Tricase
  - A.O. Universitaria S. Maria Della Misericordia Di Udine, Udine
  - Ematologia - OSPEDALE DI CIRCOLO E FONDAZIONE MACCHI, Varese